CLINICAL TRIAL: NCT04563390
Title: Effectiveness of a Projection-based Augmented Reality Exposure System in Treating Cockroach Phobia. A Randomized Controlled Trial
Brief Title: Effectiveness of a Projection-based Augmented Reality Exposure System in Treating Cockroach Phobia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TERA-P EY CP
Record Dates: First submitted 2020-09-16; First posted 2020-09-24 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Specific Phobia
Keywords: Specific phobia; Cockroach phobia; Exposure therapy; In vivo exposure; Projection-Based augmented reality therapy; Randomized Controlled Trial
MeSH Terms: conditions — Phobia, Specific

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with two treatment conditions and one WL control condition.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Projection-based augmented reality exposure therapy (Experimental): Intervention group that receives the projection-based augmented reality to carry out the exposure therapy for cockroach phobia.
  Interventions: Behavioral: Projection-based augmented reality exposure therapy (P-ARET).
- In vivo exposure (Experimental): Intervention group that receives traditional in vivo exposure therapy for cockroach phobia.
  Interventions: Behavioral: In vivo exposure therapy
- WL Control (No Intervention): Waiting list control group.

INTERVENTIONS:
Behavioral: Projection-based augmented reality exposure therapy (P-ARET). — The intervention will be based on exposure therapy to cockroaches using P-ARET. The treatment will follow the guidelines of the "one-session treatment" (OST). Main components: Psychoeducation, Exposure to the feared object (cockroach), modeling (the therapist will interact with the phobic stimulus first and if possible, the patient will follow the same steps), cognitive challenge, and reinforcement and relapse prevention.
  Arms: Projection-based augmented reality exposure therapy
Behavioral: In vivo exposure therapy — The intervention will be based on traditional in vivo exposure therapy to real cockroaches. The treatment will follow the guidelines of the "one-session treatment" (OST). Main components: Psychoeducation, Exposure to the feared object (cockroach), modeling (the therapist will interact with the phobic stimulus first and if possible, the patient will follow the same steps), cognitive challenge, and reinforcement and relapse prevention.
  Arms: In vivo exposure

SUMMARY:
The main aim of this study is to validate and test the clinical effectiveness of the projection-based augmented reality system in cockroach phobia exposure therapy through an RCT that includes three conditions: (i) projection-based augmented reality therapy, (ii) usual treatment (in vivo exposure), (iii) waiting list control. In addition, it is intended to analyze the potential of the eye-tracking technology as a tool for evaluating the clinical effectiveness in cockroach phobia treatment.

DETAILED DESCRIPTION:
The measurement of attentional biases as a clinical evaluation tool in anxiety disorders is presented as a valuable instrument capable of evaluating changes in the automatic cognitive processes that are involved in their maintenance. However, the variability between the different methodologies used for its measurement has produced a lack of empirical consistency that supports the use of this tool with a clinical purpose. The appearance and implementation of eye tracking technology in experimental studies has made it possible to overcome this problem. Despite this, to our knowledge, there are still no studies that implement this technology in the clinical field as a tool for evaluating therapeutic effectiveness.

Specific phobia is the anxiety disorder with the highest prevalence and, specifically the animal subtype, is one of the most prevalent (3.8%), producing a significant interference and high comorbidity. Despite that in vivo exposure therapy is the treatment of choice for specific phobia, the high dropout rates and difficulties in its application pose major limitations for its therapeutic implementation. The emergence of technologies such as augmented reality (AR) has made it possible to overcome these barriers, offering new ways of applying exposure therapy. AR technology offers the capacity to interact with the stimulus in the real world, facilitating the therapeutic process and the generalization of its results. Some studies have tested the effectivity and efficacy of the AR technology in small animals exposure treatment revealing promising results. However, these studies used a version of AR that requires the use of a device placed on the participant's head (HDM-Head Mounted Display) which can cause dizziness and back pain in some participants and limits the therapist-patient communication. An improved version of the AR system based on projection helps to solve this problem, allowing a more natural interaction with the stimulus and the therapist and greater comfort. The preliminary efficacy of this system has been tested in a case study but, so far, there is no RCT evaluating the efficacy of this AR system. Therefore, in this work two objectives are pursued, firstly, to test and validate a projection-based AR system in the phobia of cockroaches treatment and, secondly, to evaluate the clinical potential of the eye-tracking technology as a specific measure to assess changes in cognitive processes.

The Randomized Clinical Trial (RCT) will be conducted following the Consolidated Standards of Reporting Trials (CONSORT: http://www.consort-statement.org) and the SPIRIT guidelines (Standard Protocol Items: Recommendations for Intervention Trials). Participants (N=96) will be randomized into three groups (after receiving a SP diagnosis - DSM-5): 1) Projection-based augmented reality therapy (P-ARET); 2) In vivo Exposure therapy (IVET); and 3) a waiting list control group (WL). Participants in the WL will be randomly assigned to one of the two treatment conditions after spending time on the waiting list (1 week) for ethical reasons. Outcome measures will be assessed at baseline, post-treatment and 1-, 6-, and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Meeting DSM-5 diagnostic criteria for SP (animal subtype) to cockroaches
* Having a minimum of six-month duration of the phobia
* Sign an informed consent
* Presenting a score of at least 4 on the fear and avoidance scales of the diagnostic interview applied

Exclusion Criteria:

* Presence of another severe mental disorder that requires immediate attention
* Having current alcohol or drug dependence or abuse, psychosis or severe organic illness
* Currently being treated in a similar treatment program
* Being capable of inserting their hands in a plastic container with a cockroach (during the behavioral test)
* Receiving other psychological treatment during the study for cockroach phobia
* Start receiving pharmacological treatment during the study (or in case of being already taking them, change the drug or dose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Behavioral Avoidance Test (BAT; adapted from Öst, Salkovskis, & Hellström's, 1991) | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months).
  Patients will be confronted to a real cockroach and they will be encouraged to get closer and interact with the stimulus as much as they can. The anxiety level (0-10), distance and level of interaction with the animal will be registered and evaluated on a scale ranging from 0 (the participant does not enter the room) to 12 (the participant interacts with the cockroach).

SECONDARY OUTCOMES:
Change in attentional biases | Baseline and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months)
  An eye-tracking attentional task has been specifically designed for this project. This task evaluates the attentional bias toward cockroaches in terms of time, gaze direction and visual scanning pattern and can reveal changes in attentional bias after the treatment compared to the start
Change in Fear of Cockroaches Questionnaire (adapted from Fear of Spiders Questionnaire; FSQ, Szymanski & O'Donohue, 1995) | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months).
  This questionnaire assesses the level of fear to cockroaches. It has 18 items evaluated in a scale ranging from 1 (nothing) to 7 (very much).
Change in Cockroach Phobia Beliefs Questionnaire (SBQ; adapted from Spider Phobia Beliefs Questionnaire; SBQ, Arntz, Lavy, van der Berg & van Rijssoort, 1993). | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months).
  This questionnaire assesses two different constructs, namely catastrophic beliefs about cockroaches and beliefs about the patient's own ability to cope with a cockroach. It has 48 items evaluated in a scale ranging from 0 (I don´t believe so) to 100 (I´m convinced of it).
Change in Fear and Avoidance Scales (adapted from Marks & Mathews, 1979). | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months).
  This instrument assesses the level of fear and avoidance to the feared stimulus (i. e., cockroaches), ranged from 0 (nothing) to 10 (very much). It evaluates target behavior, negative thoughts and modulators.
Change in Patient's Improvement Scale (adapted from the Clinical Global Impression scale; CGI, Guy, 1976). | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months).
  This instrument evaluates the degree of improvement of the patient' symptoms after the treatment compared to the start. It is ranged from 1 (much worse) and 7 (much better).

OTHER OUTCOMES:
Change in Anxiety Disorders Interview Schedule for DSM-IV-TR (ADIS-IV) - Specific Phobia | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months).
  Diagnostic interview for specific phobia based on DSM-IV-TR criteria.
Change in Disgust Propensity and Sensitivity Scale-Revised-12 (DPSS-R-12; Sandín et al., 2008) | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months).
  This questionnaire includes two subscales that measure propensity to disgust and sensitivity to disgust. It contains 12 items ranged from 1 (never) to 5 (always).
Change in The Clinician Severity Scale (adapted from Di Nardo, Brown & Barlow, 1994) | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months).
  This instrument assesses the severity of symptoms evaluated by the clinician and the scale ranged from 0 (absent) to 8 (very severe).
Change in Scale of expectation and satisfaction with the treatment (adapted from Borkovec y Nau, 1972) | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months).
  This instrument contains 6 items ranged from 0 (nothing) to 10 (very much) assessing the patient's opinions about the treatment, focusing on their expectations and degree of satisfaction.
Change in Beck Depression Inventory 2nd edition (BDI-II; Beck, Steer, Brown, 1996; Spanish validation from Sanz, Navarro y Vázquez, 2003) | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months).
  This instrument assesses the existence and severity of symptoms of depression following the DSM-IV criteria. The BDI-II is a self report instrument that contains 21 items ranged from 0 to 3.
Change in State-Trait Anxiety Inventory (adapted from Laux, Glanzmann, Schaffner, & Spielberger, 1981) | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months).
  This instrument includes two scales designed to assess state and trait anxiety respectively. Each scale contains 20 items ranged from 0 (nothing/rarely) to 3 (very much/always).

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Quero, Psychology, Principal Investigator — Universitat Jaume I
Locations (1):
- Universitat Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Yes
Authors declare that due to ethical and legal reasons according to the preservation of the privacy of the participants the data from the clinical trial will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Wrzesien, M., Botella, C., Bretón-López, J., del Río González, E., Burkhardt, J. M., Alcañiz, M., & Pérez-Ara, M. Á. (2015). Treating small animal phobias using a projective-augmented reality system: A single-case study. Computers in Human Behavior, 49, 343-353.
- [Background] Tobon, J. I., Ouimet, A. J., & Dozois, D. J. (2011). Attentional bias in anxiety disorders following cognitive behavioral treatment. Journal of Cognitive Psychotherapy, 25(2), 114-129.
- [Result] Botella C, Perez-Ara MA, Breton-Lopez J, Quero S, Garcia-Palacios A, Banos RM. In Vivo versus Augmented Reality Exposure in the Treatment of Small Animal Phobia: A Randomized Controlled Trial. PLoS One. 2016 Feb 17;11(2):e0148237. doi: 10.1371/journal.pone.0148237. eCollection 2016. PMID 26886423
- [Result] Thorpe SJ, Salkovskis PM. The effect of one-session treatment for spider phobia on attentional bias and beliefs. Br J Clin Psychol. 1997 May;36(2):225-41. doi: 10.1111/j.2044-8260.1997.tb01409.x. PMID 9167863
- [Derived] Grimaldos J, Breton-Lopez J, Palau-Batet M, Diaz-Sanahuja L, Quero S. Effectiveness of a projection-based augmented reality exposure system in treating cockroach phobia: study protocol of a randomised controlled trial. BMJ Open. 2023 May 19;13(5):e069025. doi: 10.1136/bmjopen-2022-069025. PMID 37208132